CLINICAL TRIAL: NCT04674605
Title: A Prospective Cohort Study Of Myasthenia Gravis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Fei Xiao, Prof.Fei Xiao, First Affiliated Hospital of Chongqing Medical University
Other Study IDs: 2020-382
Record Dates: First submitted 2020-12-14; First posted 2020-12-19 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Myasthenia Gravis; Myasthenia Gravis Crisis
Keywords: Myasthenia Gravis; Prognostic prediction
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ocular myasthenia gravis
  Interventions: Device: biomarkers
- generalized myasthenia gravis
  Interventions: Device: biomarkers

INTERVENTIONS:
Device: biomarkers — biomarkers

SUMMARY:
The average annual incidence of Myasthenia gravis is up to (8.0-20.0) / 100,000 people. Myasthenia gravis is an acquired autoimmune disease. All skeletal muscles of patients may be involved. When ocular muscles are involved, ptosis, diplopia and other symptoms may occur. When the laryngopharyngeal muscles are involved, the patient may develop dysarthria, dysphagia and other symptoms. However, when the respiratory muscles are involved, patients will have difficulty in breathing, and some patients may develope myasthenia crisis, and artificial assisted respiratory therapy is often needed.

This study is a prospective observational study, in which patients are continuously enrolled, basic information of patients is collected, and biological samples are collected. The purpose of this study is to improve the diagnosis and prognosis of myasthenia gravis patients.

ELIGIBILITY:
Inclusion Criteria:

* Meeting the diagnosis of myasthenia gravis

Exclusion Criteria:

* Malignant tumor or other serious chronic disease

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chinese
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-12-31 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Myasthenia gravis foundation of America post intervention status | 3 years
  Complete Stable Remission (CSR) Pharmacologic Remission (PR) Minimal Manifestations (MM) Change in Status: Improved (I) Unchanged (U) Worse (W) Exacerbation (E) Died of MG (D of MG)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, YuZhong District

IPD SHARING:
Plan to Share IPD: Undecided